CLINICAL TRIAL: NCT01245439
Title: Local Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of Tocilizumab in Patients With Active Rheumatoid Arthritis on Background Non-biologic DMARDs Who Have an Inadequate Response to Current Non-biologic DMARD
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25095
Record Dates: First submitted 2010-11-17; First posted 2010-11-22 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg intravenous infusion every 4 weeks for a total of 6 infusions

SUMMARY:
This open-label study will evaluate the safety, tolerability and efficacy of RoActemra/Actemra (tocilizumab) in patients with moderate to severe active rheumatoid arthritis (RA) on background non-biologic DMARDs who have an inadequate response to current non-biologic DMARDs. Patients will receive 8 mg/kg RoActemra/Actemra as an intravenous infusion every 24 weeks for a total of 6 infusions. The anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Moderate to severe active rheumatoid arthritis (DAS28>/=3.2) of >/=6 months duration
* Body weight </=150 kg
* Patients are on one or more non-biologic DMARDs at a stable dose for a period >/=8 weeks prior to study treatment
* Patients with inadequate clinical response to a stable dose of non-biologic DMARD

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization
* Rheumatic autoimmune disease other than rheumatoid arthritis, including systemic lupus erythematosus, mixed connective tissue disease, scleroderma, polymyositis, or significant systemic involvement secondary to rheumatoid arthritis
* History of or current inflammatory joint disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Turkey (Türkiye) (14):
  - Adana
  - Ankara
  - Aydin
  - Bursa
  - Denizli
  - Elâzığ
  - Gaziantep
  - Istanbul
  - Izmir
  - İzmit
  - Konya
  - Manisa
  - Samsun
  - Sivas

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 Milligrams Per Kilogram (mg/kg): Participants received tocilizumab 8 mg/kg (not more than 800 mg) intravenous infusion every 4 weeks for 24 weeks (total of 6 infusions). Participants received tocilizumab monotherapy if they were not tolerating current Disease-modifying antirheumatic drugs (DMARDs) and those who tolerated DMARDs were on the same regimen of tocilizumab in combination with their non-biologic DMARDs.
Period: Overall Study
Arm/Group | Tocilizumab 8 Milligrams Per Kilogram (mg/kg)
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population consisted of all participants included in the study who received at least one dose of study medication.
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg (not more than 800 mg) intravenous infusion every 4 weeks for 24 weeks (total of 6 infusions). Participants received tocilizumab monotherapy if they were not tolerating current DMARDs and those who tolerated DMARDs were on the same regimen of tocilizumab in combination with their non-biologic DMARDs.
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Safety: Percentage of Participants With Treatment Emergent Adverse /Serious Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. An AE was considered treatment emergent if the date of onset of the AE was on or after the date of first dose of study medication. AEs of special interest included Major Adverse Cardiovascular Events (MACE) (including strokes), infections, and infusion reactions. An AE was considered an infection if the preferred term was in the predefined infection AE group term. A serious infection was an infection which was also considered as an AE. An AE was considered an infusion reaction if it occurred during or within 24 hours of an infusion.
Time Frame: 24 weeks
Population: The safety population consisted of all participants included in the study who received at least one dose of study medication and who had at least one post-baseline assessment of safety (that is post-baseline laboratory data, vital signs or adverse events).
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
percentage of participants
  AEs | 90.8
  SAEs | 9.2
  AEs of special interest | 52.3

2. Secondary Outcome: Percentage of Participants With All-Cause Discontinuation
Description: Participants who discontinued treatment due to any reason were included in this measure.
Time Frame: 24 weeks
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
percentage of participants | 0.0

3. Secondary Outcome: Number of Participants With Alanine Transaminase (ALT) and Asapartate Transaminase (AST) Elevations of Greater Than (>) 1.5 Upper Limit of Normal (ULN), >3 ULN and > 5 ULN
Description: Elevations in ALT and AST could indicate hepatotoxicity.
Time Frame: Screening (Visit 1), Weeks 0 (Visit 2), 4 (Visit 3), 8 (Visit 4), 12 (Visit 5), 16 (Visit 6), 20 (Visit 7) and 24 (Visit 8)
Population: Safety population
Measure: Number; unit: participants
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg (not more than 800 mg) intravenous infusion every 4 weeks for 24 weeks (total of 6 infusions). Participants received tocilizumab monotherapy if they were not tolerating current Disease-modifying antirheumatic drugs (DMARDs) and those who tolerated DMARDs were on the same regimen of tocilizumab in combination with their non-biologic DMARDs.
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
participants
  ALT (Visit 1) >1.5 ULN | 1
  ALT (Visit 1) >3 ULN | 0
  ALT (Visit 1) >5 ULN | 0
  ALT (Visit 2) >1.5 ULN | 2
  ALT (Visit 2) >3 ULN | 0
  ALT (Visit 2) >5 ULN | 0
  ALT (Visit 3) >1.5 ULN | 8
  ALT (Visit 3) >3 ULN | 1
  ALT (Visit 3) >5 ULN | 0
  ALT (Visit 4) >1.5 ULN | 5
  ALT (Visit 4) >3 ULN | 1
  ALT (Visit 4) >5 ULN | 0
  ALT (Visit 5) >1.5 ULN | 7
  ALT (Visit 5) >3 ULN | 0
  ALT (Visit 5) >5 ULN | 0
  ALT (Visit 6) >1.5 ULN | 3
  ALT (Visit 6) >3 ULN | 0
  ALT (Visit 6) >5 ULN | 0
  ALT (Visit 7) >1.5 ULN | 10
  ALT (Visit 7) >3 ULN | 0
  ALT (Visit 7) >5 ULN | 0
  ALT (Visit 8) >1.5 ULN | 12
  ALT (Visit 8) >3 ULN | 1
  ALT (Visit 8) >5 ULN | 1
  AST (Visit 1) >1.5 ULN | 0
  AST (Visit 1) >3 ULN | 0
  AST (Visit 1) >5 ULN | 0
  AST (Visit 2) >1.5 ULN | 0
  AST (Visit 2) >3 ULN | 0
  AST (Visit 2) >5 ULN | 0
  AST (Visit 3) >1.5 ULN | 0
  AST (Visit 3) >3 ULN | 0
  AST (Visit 3) >5 ULN | 0
  AST (Visit 4) >1.5 ULN | 1
  AST (Visit 4) >3 ULN | 0
  AST (Visit 4) >5 ULN | 0
  AST (Visit 5) >1.5 ULN | 1
  AST (Visit 5) >3 ULN | 0
  AST (Visit 5) >5 ULN | 0
  AST (Visit 6) >1.5 ULN | 1
  AST (Visit 6) >3 ULN | 0
  AST (Visit 6) >5 ULN | 0
  AST (Visit 7) >1.5 ULN | 5
  AST (Visit 7) >3 ULN | 0
  AST (Visit 7) >5 ULN | 0
  AST (Visit 8) >1.5 ULN | 1
  AST (Visit 8) >3 ULN | 1
  AST (Visit 8) >5 ULN | 1

4. Secondary Outcome: Percentage of Participants With ALT and AST Elevations of >1.5 ULN, >3 ULN and > 5 ULN
Description: Elevations in ALT and AST could indicate hepatotoxicity.
Time Frame: as for outcome 3
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
percentage of participants
  ALT (Visit 1) 1.5 ULN | 1.5
  ALT (Visit 1) >3 ULN | 0.0
  ALT (Visit 1) >5 ULN | 0.0
  ALT (Visit 2) >1.5 ULN | 3.1
  ALT (Visit 2) >3 ULN | 0.0
  ALT (Visit 2) >5 ULN | 0.0
  ALT (Visit 3) >1.5 ULN | 12.3
  ALT (Visit 3) >3 ULN | 1.5
  ALT (Visit 3)> 5 ULN | 0.0
  ALT (Visit 4) >1.5 ULN | 7.7
  ALT (Visit 4) >3 ULN | 1.5
  ALT (Visit 4)> 5 ULN | 0.0
  ALT (Visit 5) >1.5 ULN | 10.8
  ALT (Visit 5) >3 ULN | 0.0
  ALT (Visit 5) >5 ULN | 0.0
  ALT (Visit 6)> 1.5 ULN | 4.6
  ALT (Visit 6) >3 ULN | 0.0
  ALT (Visit 6) >5 ULN | 0.0
  ALT (Visit 7) > 1.5 ULN | 15.4
  ALT (Visit 7) >3 ULN | 0.0
  ALT (Visit 7) >5 ULN | 0.0
  ALT (Visit 8) >1.5 ULN | 18.5
  ALT (Visit 8) >3 ULN | 1.5
  ALT (Visit 8) >5 ULN | 1.5
  AST (Visit 1) >1.5 ULN | 0.0
  AST (Visit 1) >3 ULN | 0.0
  AST (Visit 1) >5 ULN | 0.0
  AST (Visit 2) >1.5 ULN | 0.0
  AST (Visit 2) >3 ULN | 0.0
  AST (Visit 2) >5 ULN | 0.0
  AST (Visit 3) >1.5 ULN | 0.0
  AST (Visit 3) >3 ULN | 0.0
  AST (Visit 3) >5 ULN | 0.0
  AST (Visit 4) >1.5 ULN | 4
  AST (Visit 4) >3 ULN | 0.0
  AST (Visit 4) >5 ULN | 0.0
  AST (Visit 5) >1.5 ULN | 4.2
  AST (Visit 5) >3 ULN | 0.0
  AST (Visit 5) >5 ULN | 0.0
  AST (Visit 6) >1.5 ULN | 1.5
  AST (Visit 6) >3 ULN | 0.0
  AST (Visit 6) >5 ULN | 0.0
  AST (Visit 7) >1.5 ULN | 7.7
  AST (Visit 7) >3 ULN | 0.0
  AST (Visit 7) >5 ULN | 0.0
  AST (Visit 8) >1.5 ULN | 1.5
  AST (Visit 8) >3 ULN | 1.5
  AST (Visit 8) >5 ULN | 1.5

5. Secondary Outcome: Percentage of Participants With Serious Infections
Description: A serious infection was an infection which was also considered as an SAE. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly
Time Frame: Weeks 4 (Visit 3), 8 (Visit 4), and 16 (Visit 6)
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
percentage of participants
  Visit 3 | 1.5
  Visit 4 | 1.5
  Visit 6 | 1.5

6. Secondary Outcome: Number of Participants With Serious Infections
Description: as for outcome 5
Time Frame: Weeks 4 (Visit 3), 8 (Visit 4), and 16 (Visit 6)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
participants
  Visit 3 | 1
  Visit 4 | 1
  Visit 6 | 1

7. Secondary Outcome: Change From Baseline to Highest Values for ALT and AST
Description: Elevations in ALT and AST could indicate hepatotoxicity. These enzymes were measured as International Units per Liter (IU/L). The change from baseline was calculated as: baseline value minus the highest value observed post-baseline for each enzyme.
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
IU/L
  ALT | 28.9 (25.2)
  AST | 21.3 (37.9)

8. Secondary Outcome: Change From Baseline to Highest Values for Low Density Lipoprotein (LDL) and Total Cholesterol
Description: Elevations in LDL and total cholesterol could lead to heart disease. The change from baseline was calculated as: baseline value minus the highest value observed post-baseline and was measured as milligrams per deciliter (mg/dL).
Time Frame: Baseline to Week 24
Population: Safety population; number of participants analyzed signifies participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 61
mg/dL
  LDL | 29.1 (27.2)
  Total Cholesterol | 39.8 (29.7)

9. Secondary Outcome: Change From Baseline to Lowest Value for Absolute Neutrophil Count (ANC)
Description: ANC is a measure of number of neutrophil granulocytes. An ANC less than 500 cells per microliter (cells/µL) is defined as neutropenia and significantly increases risk of infection. The change from baseline was calculated as: baseline value minus the highest value observed post-baseline. ANC was measured in cells/µL.
Time Frame: Baseline to Week 24
Population: Safety population
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
cells/µL | -3.04 (2.5)

10. Secondary Outcome: Number of Participants With Elevations in Lipids According to Adult Treatment Panel (ATP) III Guidelines
Description: ATP III guidelines classify LDL cholesterol >160 mg/dL, Total cholesterol >240 mg/dL, High Density Lipoprotein (HDL) >60 mg/dL and Triglycerides (TG) >199 as elevated.
Time Frame: Screening (Visit 1), Weeks 0 (Visit 2), 4 (Visit 3), 8 (Visit 4),12 (Visit 5),16 (Visit 6), 20 (Visit 7) and 24 (Visit 8)
Population: Safety population; Number (n) equals (=) number of participants analyzed at the specified visit for the given parameter.
Measure: Number; unit: participants
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg (not more than 800 mg) intravenous infusion every 4 weeks for 24 weeks (total of 6 infusions). Participants received tocilizumab monotherapy if they were not tolerating current (DMARDs and those who tolerated DMARDs were on the same regimen of tocilizumab in combination with their non-biologic DMARDs.
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
participants
  Visit 1 LDL >160 (n=62) | 3
  Visit 1 Total Cholesterol >240 (n=62) | 5
  Visit 1 HDL >60 (n=63) | 20
  Visit 1 TG>199 (n=63) | 7
  Visit 2 LDL >160 (n=57) | 1
  Visit 2 Total Cholesterol >240 (n=59) | 3
  Visit 2 HDL >60 (n=62) | 17
  Visit 2 TG>199 (n=59) | 9
  Visit 3 LDL >160 (n=60) | 6
  Visit 3 Total Cholesterol >240 (n=64) | 7
  Visit 3 HDL >60 (n=62) | 25
  Visit 3 TG>199 (n=63) | 14
  Visit 4 LDL >160 (n=55) | 5
  Visit 4 Total Cholesterol >240 (n=61) | 11
  Visit 4 HDL >60 (n=58) | 24
  Visit 4 TG>199 (n=58) | 12
  Visit 5 LDL >160 (n=62) | 7
  Visit 5 Total Cholesterol >240 (n=63) | 10
  Visit 5 HDL >60 (n=63) | 29
  Visit 5 TG>199 (n=63) | 11
  Visit 6 LDL >160 (n=59) | 5
  Visit 6 Total Cholesterol >240 (n=62) | 10
  Visit 6 HDL >60 (n=62) | 29
  Visit 6 TG>199 (n=62) | 13
  Visit 7 LDL >160 (n=62) | 5
  Visit 7 Total Cholesterol >240 (n=62) | 7
  Visit 7 HDL >60 (n=62) | 26
  Visit 7 TG>199 (n=62) | 10
  Visit 8 LDL >160 (n=61) | 8
  Visit 8 Total Cholesterol >240 (n=62) | 12
  Visit 8 HDL >60 (n=62) | 30
  Visit 8 TG>199 (n=61) | 8

11. Secondary Outcome: Percentage of Participants With Elevations in Lipids According to ATP III Guidelines
Description: ATP III guidelines classify LDL cholesterol >160 mg/dL , Total cholesterol >240 mg/dL, HDL >60 mg/dL and TG >199 as elevated.
Time Frame: as for outcome 3
Population: Safety population; n = number of participants analyzed at the specified visit for the given parameter.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
percentage of participants
  Visit 1 LDL >160 (n=62) | 4.8
  Visit 1 Total Cholesterol >240 (n=62) | 8.1
  Visit 1 HDL >60 (n=63) | 31.7
  Visit 1 TG>199 (n=63) | 11.1
  Visit 2 LDL >160 (n=57) | 1.8
  Visit 2 Total Cholesterol >240 (n=59) | 5.1
  Visit 2 HDL >60 (n=62) | 27.4
  Visit 2 TG>199 (n=59) | 15.3
  Visit 3 LDL >160 (n=60) | 10.0
  Visit 3 Total Cholesterol >240 (n=64) | 10.9
  Visit 3 HDL >60 (n=62) | 40.3
  Visit 3 TG>199 (n=63) | 22.2
  Visit 4 LDL >160 (n=55) | 7.3
  Visit 4 Total Cholesterol >240 (n=61) | 18.0
  Visit 4 HDL >60 (n=58) | 41.4
  Visit 4 TG>199 (n=58) | 20.7
  Visit 5 LDL >160 (n=62) | 11.3
  Visit 5 Total Cholesterol >240 (n=63) | 15.9
  Visit 5 HDL >60 (n=63) | 46.0
  Visit 5 TG>199 (n=63) | 17.5
  Visit 6 LDL >160 (n=59) | 8.5
  Visit 6 Total Cholesterol >240 (n=62) | 16.1
  Visit 6 HDL >60 (n=62) | 46.8
  Visit 6 TG>199 (n=62) | 21.0
  Visit 7 LDL >160 (n=62) | 8.1
  Visit 7 Total Cholesterol >240 (n=62) | 11.3
  Visit 7 HDL >60 (n=62) | 41.9
  Visit 7 TG>199 (n=62) | 16.1
  Visit 8 LDL >160 (n=61) | 13.1
  Visit 8 Total Cholesterol >240 (n=62) | 19.4
  Visit 8 HDL >60 (n=62) | 48.4
  Visit 8 TG>199 (n=61) | 13.1

12. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful Improvement in Disease Activity Score 28 (DAS28) At Every Visit
Description: The DAS28 is a combined index for measuring disease activity in Rheumatoid Arthritis (RA). The index includes swollen and tender joint counts, acute phase response, and general health status. The DAS28, which uses a 28 joint count, is derived from the original DAS. The index is calculated using the following formula:
  DAS28 = 0.56 x (TJC28)^0.5 + 0.28 x (SJC28)^0.5 + 0.70 x In(ESR) + 0.014 x GH Where TJC28 = tender joint count on 28 joints, SJCz8 = swollen joint count on 28 joints, ın = natural log, ESR = erythrocyte sedimentation rate and GH = general health (participant's global assessment of disease activity). DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A score of less than (<) 2.6 represents clinical remission, a score of: <3.2 represents low disease activity (LDA), and a score of > 5.1 represents severe disease. A reduction from previous visit of at least 1.2 units in DAS28 is considered to be a clinically meaningful improvement.
Time Frame: as for outcome 3
Population: Intent- to- Treat (ITT) Population: all enrolled participants who received at least one dose of study medication. Number of participants analyzed = participants who were evaluable for this outcome and n = participants who were evaluable for specified category
Measure: Number; unit: participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
participants
  Visit 1 - Visit 2 (n=55) | 0
  Visit 2 - Visit 3 (n=55) | 48
  Visit 3 - Visit 4 (n=54) | 18
  Visit 4 - Visit 5 (n=53) | 7
  Visit 5 - Visit 6 (n=54) | 2
  Visit 6 - Visit 7 (n=53) | 4
  Visit 7 - Visit 8 (n=53) | 1

13. Secondary Outcome: Percentage of Participants Who Achieved Clinically Meaningful Improvement in DAS28 At Every Visit
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen and tender joint counts, acute phase response, and general health status. The DAS28, which uses a 28 joint count, is derived from the original DAS. The index is calculated using the following formula:
  DAS28 = 0.56 x (TJC28)^0.5 + 0.28 x (SJC28)^0.5 + 0.70 x In(ESR) + 0.014 x GH Where TJC28 = tender joint count on 28 joints, SJCz8 = swollen joint count on 28 joints, ın = natural log, ESR = erythrocyte sedimentation rate and GH = general health (participant's global assessment of disease activity). DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A score of < 2.6 represents clinical remission, a score of: < 3.2 represents LDA, and a score of > 5.1 represents severe disease. A reduction of at least 1.2 units from previous visit in DAS28 is considered to be a clinically meaningful improvement.
Time Frame: as for outcome 10
Population: ITT Population; Number of participants analyzed = participants who were evaluable for this outcome and n = participants who were evaluable for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
percentage of participants
  Visit 1 - Visit 2 (n=55) | 0.0
  Visit 2 - Visit 3 (n=55) | 87.3
  Visit 3 - Visit 4 (n=54) | 33.3
  Visit 4 - Visit 5 (n=53) | 13.2
  Visit 5 - Visit 6 (n=54) | 3.7
  Visit 6 - Visit 7 (n=53) | 7.5
  Visit 7 - Visit 8 (n=53) | 1.9

14. Secondary Outcome: Number of Participants Who Achieved LDA By Visit
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen and tender joint counts, acute phase response, and general health status. The DAS28, which uses a 28 joint count, is derived from the original DAS. The index is calculated using the following formula:
  DAS28 = 0.56 x (TJC28)^0.5 + 0.28 x (SJC28)^0.5 + 0.70 x In(ESR) + 0.014 x GH Where TJC28 = tender joint count on 28 joints, SJCz8 = swollen joint count on 28 joints, ın = natural log, ESR = erythrocyte sedimentation rate and GH = general health (participant's global assessment of disease activity). DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A score of < 2.6 represents clinical remission, a score of: <3.2 represents LDA, and a score of > 5.1 represents severe disease. A reduction of at least 1.2 units from previous visit in DAS28 is considered to be a clinically meaningful improvement.
Time Frame: as for outcome 3
Population: ITT Population; Number of participants analyzed = participants who were evaluable for this outcome and n = number of participants who were evaluable for the specified category.
Measure: Number; unit: participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
participants
  Visit 1 (n=60) | 0
  Visit 2 (n=58) | 1
  Visit 3 (n=57) | 32
  Visit 4 (n=56) | 45
  Visit 5 (n=57) | 48
  Visit 6 (n=57) | 50
  Visit 7 (n=54) | 51
  Visit 8 (n=60) | 55

15. Secondary Outcome: Percentage of Participants Who Achieved LDA By Visit
Description: TThe DAS28 is a combined index for measuring disease activity in RA. The index includes swollen and tender joint counts, acute phase response, and general health status. The DAS28, which uses a 28 joint count, is derived from the original DAS. The index is calculated using the following formula:
  DAS28 = 0.56 x (TJC28)^0.5 + 0.28 x (SJC28)^0.5 + 0.70 x In(ESR) + 0.014 x GH Where TJC28 = tender joint count on 28 joints, SJCz8 = swollen joint count on 28 joints, ın = natural log, ESR = erythrocyte sedimentation rate and GH = general health (participant's global assessment of disease activity). DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A score of < 2.6 represents clinical remission, a score of: <3.2 represents LDA, and a score of > 5.1 represents severe disease. A reduction of at least 1.2 units from previous visit in DAS28 is considered to be a clinically meaningful improvement.
Time Frame: as for outcome 3
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
percentage of participants
  Visit 1 (n=60) | 0.0
  Visit 2 (n=58) | 1.7
  Visit 3 (n=57) | 56.1
  Visit 4 (n=56) | 80.4
  Visit 5 (n=57) | 84.2
  Visit 6 (n=57) | 87.7
  Visit 7 (n=54) | 94.4
  Visit 8 (n=60) | 91.7

16. Secondary Outcome: Time to LDA (DAS28 ) Based on First Visit When LDA Was Observed
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen and tender joint counts, acute phase response, and general health status. The DAS28, which uses a 28 joint count, is derived from the original DAS. The index is calculated using the following formula:
  DAS28 = 0.56 x (TJC28)^0.5 + 0.28 x (SJC28)^0.5 + 0.70 x In(ESR) + 0.014 x GH Where TJC28 = tender joint count on 28 joints, SJCz8 = swollen joint count on 28 joints, ın = natural log, ESR = erythrocyte sedimentation rate and GH = general health (participant's global assessment of disease activity). DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A score of < 2.6 represents clinical remission, a score of: <3.2 LDA, and a score of > 5.1 represents severe disease. A reduction of at least 1.2 units from previous visit in DAS28 is considered to be a clinically meaningful improvement.
Time Frame: as for outcome 3
Population: ITT Population; Number of participants analyzed = participants who were evaluable for this outcome
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
Percentage of participants
  Visit 1 | 0.0
  Visit 2 | 1.7
  Visit 3 | 51.7
  Visit 4 | 28.3
  Visit 5 | 10.0
  Visit 6 | 1.7
  Visit 7 | 1.7
  Visit 8 | 1.7
  Never Acheived LDA | 3.3

17. Secondary Outcome: Number of Participants Who Achieved Remission (DAS28) By Visit
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen and tender joint counts, acute phase response, and general health status. The DAS28, which uses a 28 joint count, is derived from the original DAS. The index is calculated using the following formula:
  DAS28 = 0.56 x (TJC28)^0.5 + 0.28 x (SJC28)^0.5 + 0.70 x In(ESR) + 0.014 x GH Where TJC28 = tender joint count on 28 joints, SJCz8 = swollen joint count on 28 joints, ın = natural log, ESR = erythrocyte sedimentation rate and GH = general health (participant's global assessment of disease activity). DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A score of < 2.6 represents clinical remission, a score of: <3.2 LDA, and a score of > 5.1 represents severe disease. A reduction of at least 1.2 units in DAS28 is considered to be a clinically meaningful improvement.
Time Frame: as for outcome 3
Population: ITT population. Number of participants analyzed = participants who were evaluable for this outcome and n = participants who were evaluable for specified category
Measure: Number; unit: participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
participants
  Visit (n=60) | 0
  Visit 2 (n=58) | 0
  Visit 3 (n=57) | 24
  Visit 4 (n=56) | 35
  Visit 5 (n=57) | 43
  Visit 6 (n=57) | 46
  Visit 7 (n=54) | 45
  Visit 8 (n=60) | 51

18. Secondary Outcome: Percentage of Participants Who Achieved Remission (DAS28) At Every Visit
Description: as for outcome 17
Time Frame: as for outcome 3
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome and n = participants who were evaluable for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
percentage of participants
  Visit 1 (n=60) | 0.0
  Visit 2 (n=58) | 0.0
  Visit 3 (n=57) | 42.1
  Visit 4 (n=56) | 62.5
  Visit 5 (n=57) | 75.4
  Visit 6 (n=57) | 80.7
  Visit 7 (n=54) | 83.3
  Visit 8 (n=60) | 85.0

19. Secondary Outcome: Percentage of Participants Achieving Their First Remission Status By Visit
Description: as for outcome 17
Time Frame: Weeks 4 (Visit 3), 8 (Visit 4), 12 (Visit 5), 16 (Visit 6), 20 (Visit 7) and 24 (Visit 8)
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
Percentage of participants
  In Visit 3 | 40.0
  In Visit 4 | 25.0
  In Visit 5 | 15.0
  In Visit 6 | 5.0
  In Visit 7 | 3.3
  In Visit 8 | 3.3
  Never Achieved Remission | 8.3

20. Secondary Outcome: Disease Activity Score as Measured By DAS28 at Each Visit
Description: as for outcome 17
Time Frame: as for outcome 3
Population: ITT population. n = participants who were evaluable for specified category
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
units on a scale
  Visit 1 (n=60) | 5.6 (0.9)
  Visit 2 (n=58) | 5.6 (1.1)
  Visit 3 (n=57) | 3.1 (1.4)
  Visit 4 (n=56) | 2.3 (1.0)
  Visit 5 (n=57) | 2.0 (1.3)
  Visit 6 (n=57) | 1.8 (1.1)
  Visit 7 (n=54) | 1.7 (1.0)
  Visit 8 (n=60) | 1.6 (1.0)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Change from Visit 1 to Visit 2; Test type: Superiority or Other; p = 0.929, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Change from Visit 2 to 3; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Change from Visit 3 to Visit 4; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; Change from Visit 4 to Visit 5; Test type: Superiority or Other; p = 0.050, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; Change from Visit 5 to Visit 6; Test type: Superiority or Other; p = 0.165, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; Change from Visit 6 to Visit 7; Test type: Superiority or Other; p = 0.133, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Tocilizumab 8 mg/kg; Change from Visit 7 to Visit 8; Test type: Superiority or Other; p = 0.217, Wilcoxon Signed Rank test
Statistical Analysis 8: Comparison: Tocilizumab 8 mg/kg; Change from Visit 2 to Visit 8; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

21. Secondary Outcome: Number of Participants Who Achieved American College of Rheumatology (ACR) 20, ACR 50, ACR 70 and ACR 90 Response
Description: ACR20/50/70/90 response: greater than or equal to (≥) 20/50/70/90 percent (%) improvement in TJC; ≥20/50/70/90% improvement in SJC; and ≥20/50/70/90% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP). Improvements were assessed on the basis of prior visit.
Time Frame: Weeks 0 (Visit 2), 4 (Visit 3), 8 (Visit 4),12 (Visit 5),16 (Visit 6), 20 (Visit 7) and 24 (Visit 8)
Population: ITT population; number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
participants
  Visit 2 to Visit 3 ACR20 | 20
  Visit 2 to Visit 3 ACR50 | 12
  Visit 2 to Visit 3 ACR70 | 5
  Visit 2 to Visit 3 ACR90 | 0
  Visit 3 to Visit 4 ACR20 | 37
  Visit 3 to Visit 4 ACR50 | 25
  Visit 3 to Visit 4 ACR70 | 14
  Visit 3 to Visit 4 ACR90 | 1
  Visit 4 to Visit 5 ACR20 | 33
  Visit 4 to Visit 5 ACR50 | 26
  Visit 4 to Visit 5 ACR70 | 18
  Visit 4 to Visit 5 ACR90 | 4
  Visit 5 to Visit 6 ACR20 | 32
  Visit 5 to Visit 6 ACR50 | 26
  Visit 5 to Visit 6 ACR70 | 20
  Visit 5 to Visit 6 ACR90 | 7
  Visit 6 to Visit 7 ACR20 | 27
  Visit 6 to Visit 7 ACR50 | 23
  Visit 6 to Visit 7 ACR70 | 17
  Visit 6 to Visit 7 ACR90 | 4
  Visit 7 to Visit 8 ACR20 | 32
  Visit 7 to Visit 8 ACR50 | 28
  Visit 7 to Visit 8 ACR70 | 18
  Visit 7 to Visit 8 ACR90 | 6

22. Secondary Outcome: Percentage of Participants Who Achieved ACR 20, ACR 50, ACR 70 and ACR 90 Response
Description: ACR20/50/70/90 response: ≥ 20/50/70/90 % improvement in TJC; ≥20/50/70/90% improvement in SJC; and ≥20/50/70/90% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP). Improvements were assessed on the basis of prior visit. .
Time Frame: Weeks 0 (Visit 2), 4 (Visit 3), 8 (Visit 4),12 (Visit 5),16 (Visit 6), 20 (Visit 7) and 24 (Visit 8)
Population: ITT population; number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
Percentage of participants
  Visit 2 to Visit 3 ACR20 | 33.3
  Visit 2 to Visit 3 ACR50 | 20.0
  Visit 2 to Visit 3 ACR70 | 8.3
  Visit 2 to Visit 3 ACR90 | 0.0
  Visit 3 to Visit 4 ACR20 | 61.7
  Visit 3 to Visit 4 ACR50 | 41.7
  Visit 3 to Visit 4 ACR70 | 23.3
  Visit 3 to Visit 4 ACR90 | 1.7
  Visit 3 to Visit 5 ACR20 | 55.0
  Visit 4 to Visit 5 ACR50 | 43.3
  Visit 4 to Visit 5 ACR70 | 30.0
  Visit 4 to Visit 5 ACR90 | 6.7
  Visit 5 to Visit 6 ACR20 | 53.3
  Visit 5 to Visit 6 ACR50 | 43.3
  Visit 5 to Visit 6 ACR70 | 33.3
  Visit 5 to Visit 6 ACR90 | 11.7
  Visit 6 to Visit 7 ACR20 | 45.0
  Visit 6 to Visit 7 ACR50 | 38.3
  Visit 6 to Visit 7 ACR70 | 28.3
  Visit 6 to Visit 7 ACR90 | 6.7
  Visit 7 to Visit 8 ACR20 | 53.3
  Visit 7 to Visit 8 ACR50 | 46.7
  Visit 7 to Visit 8 ACR70 | 30.0
  Visit 7 to Visit 8 ACR90 | 10.0

23. Secondary Outcome: C-Reactive Protein Levels
Description: CRP is an inflammatory marker used to measure inflammation in RA and is measured as mg/dL.
Time Frame: as for outcome 3
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 59
mg/dL
  Visit 1 (n=59) | 3.5 (6.2)
  Visit 2 (n=53) | 2.3 (3.2)
  Visit 3 (n=53) | 1.0 (2.2)
  Visit 4 (n=58) | 0.6 (0.9)
  Visit 5 (n=57) | 0.6 (1.3)
  Visit 6 (n=58) | 1.0 (4.2)
  Visit 7 (n=52) | 0.8 (1.6)
  Visit 8 (n=58) | 0.5 (0.8)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Change from Visit 1 to Visit 2; Test type: Superiority or Other; p = 0.169, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Change from Visit 2 to Visit 3; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Change from Visit 3 to Visit 4; Test type: Superiority or Other; p = 0.053, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; Change from Visit 4 to Visit 5; Test type: Superiority or Other; p = 0.514, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; Change from Visit 5 to Visit 6; Test type: Superiority or Other; p = 0.064, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; Change from Visit 6 to Visit 7; Test type: Superiority or Other; p = 0.038, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Tocilizumab 8 mg/kg; Change from Visit 7 to Visit 8; Test type: Superiority or Other; p = 0.064, Wilcoxon Signed Rank test
Statistical Analysis 8: Comparison: Tocilizumab 8 mg/kg; Change from Visit 2 to Visit 8; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

24. Secondary Outcome: Erythrocyte Sedimentation Rate
Description: ESR is an inflammatory marker used to measure inflammation in RA and is measured as millimeters per hour (mm/hr).
Time Frame: as for outcome 3
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 60
mm/hr
  Visit 1 (n=60) | 35.4 (22.9)
  Visit 2 (n=58) | 36.4 (24.1)
  Visit 3 (n=57) | 12.3 (13.3)
  Visit 4 (n=56) | 8.0 (9.3)
  Visit 5 (n=58) | 7.8 (9.4)
  Visit 6 (n=57) | 7.8 (8.2)
  Visit 7 (n=54) | 6.3 (5.4)
  Visit 8 (n=60) | 8.6 (13.8)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Change from Visit 1 to Visit 2; Test type: Superiority or Other; p = 0.981, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Change from Visit 2 to Visit 3; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Change from Visit 3 to Visit 4; Test type: Superiority or Other; p = 0.005, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; Change from Visit 4 to Visit 5; Test type: Superiority or Other; p = 0.566, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; Change from Visit 5 to Visit 6; Test type: Superiority or Other; p = 0.264, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; Change from Visit 6 to Visit 7; Test type: Superiority or Other; p = 0.126, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Tocilizumab 8 mg/kg; Change from Visit 7 to Visit 8; Test type: Superiority or Other; p = 0.779, Wilcoxon Signed Rank test
Statistical Analysis 8: Comparison: Tocilizumab 8 mg/kg; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

25. Secondary Outcome: Mean Number of Tender and Swollen Joints
Description: Participants were asked to classify 28 joints as tender or not tender and swollen or not swollen to count the total number of tender and swollen joints by visit.
Time Frame: as for outcome 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
joints
  Visit 1 TJC | 15.1 (9.6)
  Visit 1 SJC | 5.5 (4.7)
  Visit 2 TJC | 16.0 (11.5)
  Visit 2 SJC | 5.7 (5.2)
  Visit 3 TJC | 6.1 (7.4)
  Visit 3 SJC | 1.9 (3.2)
  Visit 4 TJC | 3.3 (4.8)
  Visit 4 SJC | 0.8 (1.6)
  Visit 5 TJC | 2.7 (4.7)
  Visit 5 SJC | 0.5 (1.1)
  Visit 6 TJC | 2.0 (4.4)
  Visit 6 SJC | 0.5 (1.3)
  Visit 7 TJC | 1.8 (3.2)
  Visit 7 SJC | 0.6 (1.6)
  Visit 8 TJC | 1.3 (2.6)
  Visit 8 SJC | 0.4 (1.2)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Change in Sensitive Joints Visit 1 to Visit 2; Test type: Superiority or Other; p = 0.410, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Change in Sensitive Joints from Visit 2 to Visit 3; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Change in Sensitive Joints from Visit 3 to Visit 4; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; Change in Sensitive Joints from Visit 4 to Visit 5; Test type: Superiority or Other; p = 0.021, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; Change in Sensitive Joints from Visit 5 to Visit 6; Test type: Superiority or Other; p = 0.003, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; Change in Sensitive Joints from Visit 6 to Visit7; Test type: Superiority or Other; p = 0.827, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Tocilizumab 8 mg/kg; Change in Sensitive Joints from Visit 7 to Visit 8; Test type: Superiority or Other; p = 0.093, Wilcoxon Signed Rank test
Statistical Analysis 8: Comparison: Tocilizumab 8 mg/kg; Change in Sensitive Joints from Visit 2 to Visit 8; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 9: Comparison: Tocilizumab 8 mg/kg; Change in Swollen Joints from Visit 1 to Visit 2; Test type: Superiority or Other; p = 0.792, Wilcoxon Signed Rank test
Statistical Analysis 10: Comparison: Tocilizumab 8 mg/kg; Change in Swollen Joints from Visit 2 to Visit 3; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 11: Comparison: Tocilizumab 8 mg/kg; Change in Swollen Joints from Visit 3 to Visit 4; Test type: Superiority or Other; p = 0.002, Wilcoxon Signed Rank test
Statistical Analysis 12: Comparison: Tocilizumab 8 mg/kg; Change in Swollen Joints from Visit 4 to Visit 5; Test type: Superiority or Other; p = 0.374, Wilcoxon Signed Rank test
Statistical Analysis 13: Comparison: Tocilizumab 8 mg/kg; Change in Swollen Joints from Visit 5 to Visit 6; Test type: Superiority or Other; p = 0.518, Wilcoxon Signed Rank test
Statistical Analysis 14: Comparison: Tocilizumab 8 mg/kg; Change in Swollen Joints from Visit 6 to Visit 7; Test type: Superiority or Other; p = 0.744, Wilcoxon Signed Rank test
Statistical Analysis 15: Comparison: Tocilizumab 8 mg/kg; Change in Swollen Joints from Visit 7 to Visit 8; Test type: Superiority or Other; p = 0.048, Wilcoxon Signed Rank test
Statistical Analysis 16: Comparison: Tocilizumab 8 mg/kg; Change in Swollen Joints from Visit 2 to Visit 8; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

26. Secondary Outcome: Participant's (PT) and Investigator's (IN) Assessment of Disease Activity
Description: VAS is a visual scale of 100 mm for the assessment of disease activity by participants or investigator. Disease activity/pain increases while approaching 100 mm. For the screening visit (baseline visit) there's only investigator assessment data, for other visits participant's pain assessment, participant's disease activity assessment and investigator's disease activity assessment parameters were collected.
Time Frame: as for outcome 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
mm
  Visit 1 IN | 70.1 (16.0)
  Visit 2 PT | 70.3 (17.7)
  Visit 2 IN | 68.3 (16.7)
  Visit 3 PT | 41.8 (24.7)
  Visit 3 IN | 33.3 (21.5)
  Visit 4 PT | 25.3 (20.1)
  Visit 4 IN | 20.6 (14.1)
  Visit 5 PT | 24.1 (20.6)
  Visit 5 IN | 16.9 (13.8)
  Visit 6 PT | 23.1 (21.9)
  Visit 6 IN | 16.9 (16.7)
  Visit 7 PT | 18.3 (18.6)
  Visit 7 IN | 14.9 (14.4)
  Visit 8 PT | 16.2 (17.3)
  Visit 8 IN | 12.5 (14.1)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; PT assessment Visit 2 to Visit 3; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; PT assessment Visit 3 to Visit 4; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; PT assessment Visit 4 to Visit 5; Test type: Superiority or Other; p = 0.075, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; PT assessment Visit 5 to Visit 6; Test type: Superiority or Other; p = 0.119, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; PT assessment Visit 6 to Visit 7; Test type: Superiority or Other; p = 0.007, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; PT assessment Visit 7 to Visit 8; Test type: Superiority or Other; p = 0.047, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Tocilizumab 8 mg/kg; PT assessment Visit 2 to Visit 8; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 8: Comparison: Tocilizumab 8 mg/kg; IN assessment Visit 2 to Visit 3; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 9: Comparison: Tocilizumab 8 mg/kg; IN assessment Visit 3 to Visit 4; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 10: Comparison: Tocilizumab 8 mg/kg; IN assessment Visit 4 to Visit 5; Test type: Superiority or Other; p = 0.001, Wilcoxon Signed Rank test
Statistical Analysis 11: Comparison: Tocilizumab 8 mg/kg; IN assessment Visit 5 to Visit 6; Test type: Superiority or Other; p = 0.084, Wilcoxon Signed Rank test
Statistical Analysis 12: Comparison: Tocilizumab 8 mg/kg; IN assessment Visit 6 to Visit 7; Test type: Superiority or Other; p = 0.272, Wilcoxon Signed Rank test
Statistical Analysis 13: Comparison: Tocilizumab 8 mg/kg; IN assessment Visit 7 to Visit 8; Test type: Superiority or Other; p = 0.020, Wilcoxon Signed Rank test
Statistical Analysis 14: Comparison: Tocilizumab 8 mg/kg; IN assessment Visit 2 to Visit 8; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

27. Secondary Outcome: Participant's Assessment of Pain
Description: as for outcome 26
Time Frame: Weeks 0 (Visit 2), 4 (Visit 3), 8 (Visit 4), 12 (Visit 5), 16 (Visit 6), 20 (Visit 7) and 24 (Visit 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
mm
  Visit 2 | 66.4 (20.8)
  Visit 3 | 38.8 (26.7)
  Visit 4 | 25.6 (22.6)
  Visit 5 | 22.7 (21.8)
  Visit 6 | 23.0 (23.9)
  Visit 7 | 17.8 (17.9)
  Visit 8 | 15.3 (16.5)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Change between Visit 2 to Visit 3; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Change between Visit 3 to Visit 4; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Change between Visit 4 to Visit 5; Test type: Superiority or Other; p = 0.254, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; Change between Visit 5 to Visit 6; Test type: Superiority or Other; p = 0.138, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; Change between Visit 6 to Visit 7; Test type: Superiority or Other; p = 0.002, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; Change between Visit 7 to Visit 8; Test type: Superiority or Other; p = 0.104, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Tocilizumab 8 mg/kg; Change between Visit 2 to Visit 8; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

28. Secondary Outcome: Health Assessment Questionnaire Score (General Score)
Description: The Stanford HAQ disability index is a participant completed questionnaire specific for RA. It consists of 20 questions referring to 8 component sections: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. The questionnaire was provided in validated translation into the local languages at the participating sites and was scored. Every question in each section was scored at a scale from 0 to 3 by the participant where 0 = able to perform the activity without any difficulty and 3 = unable to perform the activity. General score was calculated as an average of the 8 sections.
Time Frame: Weeks 0 (Visit 2), 4 (Visit 3), 8 (Visit 4), 12 (Visit 5), 16 (Visit 6), 20 (Visit 7) and 24 (Visit 8)
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 65
units on a scale
  Visit 2 | 1.3 (0.7)
  Visit 3 | 0.8 (0.8)
  Visit 4 | 0.6 (0.7)
  Visit 5 | 0.5 (0.7)
  Visit 6 | 0.4 (0.6)
  Visit 7 | 0.4 (0.7)
  Visit 8 | 0.4 (0.6)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Change between Visit 2 to Visit 3; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Change between Visit 3 to Visit 4; Test type: Superiority or Other; p = 0.002, Wilcoxon Signed Rank test
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Change between Visit 4 to Visit 5; Test type: Superiority or Other; p = 0.078, Wilcoxon Signed Rank test
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; Change between Visit 5 to Visit 6; Test type: Superiority or Other; p = 0.349, Wilcoxon Signed Rank test
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; Change between Visit 6 to Visit 7; Test type: Superiority or Other; p = 0.722, Wilcoxon Signed Rank test
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; Change between Visit 7 to Visit 8; Test type: Superiority or Other; p = 0.224, Wilcoxon Signed Rank test

ADVERSE EVENTS:
Time Frame: From the date of first infusion to 24 weeks
Arm/Group | Tocilizumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 11/65
Other Adverse Events (participants affected / at risk) | 45/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=65)
Hypertension, tremor, acute infusion reaction (Vascular disorders) | 1
Pneumonia (community acquired pneumonia) (Infections and infestations) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (suspected) (Infections and infestations) | 1
Vasculit (splinter hemorrhage, fingertip hemorrhage) (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Hypercholesterolaemia, Hypertriglyceridaemia, LDL-Hyperlipidaemia (Investigations) | 1
Hypertriglyceridaemia (Investigations) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Elevated levels of ALT (Investigations) | 1
Cardiac pain (angina pectoris) (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=65)
Hypercholesterolaemia (Investigations) | 11
Hypertriglyceridaemia (Investigations) | 7
Elevated ALT <45 (Hepatobiliary disorders) | 11
Elevated ALT 1.5- 3 ULN (Hepatobiliary disorders) | 14
Elevated AST <60 (Hepatobiliary disorders) | 9
Elevated AST 1.5 - 3ULN (Hepatobiliary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.